CLINICAL TRIAL: NCT02469142
Title: Use of Acellular Dermal in the Incarcerated Inguinal Hernia Tension-free Reconstructions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Xiaonan Liu, Principal Investigator, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADM001
Record Dates: First submitted 2015-01-04; First posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Incarcerated Inguinal Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADM tension-free hernia reparation (Experimental): Use ADM to repair incarcerated inguinal hernia by tension-free
  Interventions: Procedure: ADM tension-free hernia reparation
- traditional tension hernia reparation (Placebo Comparator): Just repair incarcerated inguinal hernia by nothing in tension condition

INTERVENTIONS:
Procedure: ADM tension-free hernia reparation — Use ADM as opposed to nothing to repair incarcerated inguinal hernia
  Arms: ADM tension-free hernia reparation

SUMMARY:
Incarcerated inguinal hernia is one of the common acute abdomen abdominal surgery, often prone to intestinal necrosis and acute peritonitis.Using traditional tension hernia reparation, the recurrence rate were as high as 30%. In recent years, biological materials especially acellular matrix materials (Acellular Dermal Matrix, ADM) in resisting the infection, has become a research hotspot. In the project, the investigators try to address the role of ADM in incarcerated inguinal hernia patients.

DETAILED DESCRIPTION:
observation indicator:

1. recurrence rate after operation
2. incidence rate of complications
3. postoperative hospital stay
4. hospitalization costs
5. Self-evaluation of gastroesophageal reflux symptoms and quality of life(QOL) in 6th-month, 1st-year,2nd-year,3rd-year,4th-year and 5th-year after operation

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of incarcerated hernia
* randomly select patch agreed by patients and family members

Exclusion Criteria:

* severe organ dysfunction
* No-tolerate anesthesia
* No-suitable for operation
* glucocorticoid with long-term use
* Sever intraperitoneal adhesion existed
* spirit disease patients
* automatically exit

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate after operation | ten years

CONTACTS AND LOCATIONS:
Overall Officials: xiaonan liu, MD, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China

REFERENCES:
- [Derived] Saeter AH, Fonnes S, Li S, Rosenberg J, Andresen K. Mesh versus non-mesh for emergency groin hernia repair. Cochrane Database Syst Rev. 2023 Nov 27;11(11):CD015160. doi: 10.1002/14651858.CD015160.pub2. PMID 38009575